CLINICAL TRIAL: NCT05891743
Title: Prevalence of Skin Sensitization and Dermatitis Among Epoxy-exposed Workers in the Wind Turbine Industry
Acronym: EPOXY
Status: Completed | Type: Observational
Sponsor: Siemens Gamesa Renewable Energy Blades, S.A. (Industry)
Collaborators: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: LOD_VAG_011
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Dermatitis
MeSH Terms: conditions — Dermatitis | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epoxy_Group: Workers who are exposed to epoxy handling procedures, specifically filling and lamination tasks performed by production workers, mainly in finishing areas.
  Interventions: Diagnostic Test: Patch Test
- Non_exposed: Workers from other areas unrelated to epoxy handling procedures, that will be included in the study as the non-exposed control group.
  Interventions: Diagnostic Test: Patch Test

INTERVENTIONS:
Diagnostic Test: Patch Test — The Patch Test will include the European baseline series, as well as the epoxy and isocyanate series. Additionally, specific products commonly used in the workplace, such as glues, resins, and paints, will be prepared and included in the testing.

SUMMARY:
The goal of this observational study it to learn about the prevalence of skin sensitization and dermatitis among epoxy-exposed workers in the wind turbine industry. The main question it aims to answer is:

- What is the prevalence of skin sensitization and dermatitis among workers in the wind turbine industry who are exposed to epoxy?

Participants will be asked to perform Patch Test, which is considered the Gold Standard test for identifying the cause of occupational contact allergic dermatitis.

Researchers will compare the results of the epoxy-exposed group with those of a control group comprising non-exposed workers from the same industry. This analysis will help determine if there is a higher prevalence of skin sensitization among workers exposed to epoxy.

DETAILED DESCRIPTION:
Epoxy resin systems are widely used materials in various industries due to their high mechanical, chemical, and thermal resistance. These systems are commonly employed as protective coatings, adhesives, and paints, as well as in the manufacturing of composites in the plastics industry. Epoxy components are well-known sensitizers of the skin. A high prevalence of skin sensitization and dermatitis have been reported among workers exposed to epoxy components. It is recommended to use comprehensive protective equipment when handling epoxy components. In the wind turbine industry, tasks involving epoxy handling, such as lamination and filling procedures, are frequently performed. Recent study have shown a sensitization prevalence of 8.9% among workers performing these tasks, while a previous study reported a high sensitization rate of 10.5% to epoxy resins. Despite efforts to find alternatives to epoxy resin systems and improve protective measures, the use of epoxy has increased, and some countries have implemented more stringent regulations, such as Denmark. In Portugal, there are currently no specific regulations regarding epoxy handling, and no certification is required for working with epoxy. Siemens Gamesa Renewable Energy, in Portugal, faces many skin problems among production workers, however numbers are unknown. Therefore, the main purpose of the study is to evaluate the prevalence of skin sensitization and dermatitis among epoxy-exposed workers in the wind Turbine Industry.

ELIGIBILITY:
Inclusion Criteria:

* Workers from the wind turbine industry

Exclusion Criteria:

* Pregnant females
* Workers previously diagnosed with epoxy resin sensitization

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Workers from the wind turbine industry
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Prevalence of skin sensitization. | 2-3 days
  Allergens will be applied to the participant's back using IQ Chambers® (Chemotechnique) and secured with 4fix® adhesive tape for 48 hours. Readings will be conducted on day 2-3 and, if necessary, on days 4-7, following the ESCD guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Vítor Pinheiro, MD, Principal Investigator — AIBILI-CEC (AIBILI- Clinical Trials Centre)
Locations (1):
- Siemens Gamesa Renewable Energy (SGRE), Aveiro, Soza, Portugal

REFERENCES:
- [Background] Aalto-Korte K, Pesonen M, Suuronen K. Occupational allergic contact dermatitis caused by epoxy chemicals: occupations, sensitizing products, and diagnosis. Contact Dermatitis. 2015 Dec;73(6):336-42. doi: 10.1111/cod.12445. Epub 2015 Jul 30. PMID 26230376
- [Background] Prodi A, Rui F, Fortina AB, Corradin MT, Filon FL. Occupational sensitization to epoxy resins in Northeastern Italy (1996-2010). Int J Occup Environ Health. 2015;21(1):82-7. doi: 10.1179/2049396714Y.0000000095. PMID 25633931
- [Background] Geier J, Lessmann H, Hillen U, Skudlik C, Jappe U. Sensitization to reactive diluents and hardeners in epoxy resin systems. IVDK data 2002-2011. Part II: concomitant reactions. Contact Dermatitis. 2016 Feb;74(2):94-101. doi: 10.1111/cod.12490. Epub 2015 Nov 5. PMID 26537833
- [Background] Christiansen AG, Carstensen O, Sommerlund M, Clausen PA, Bonlokke JH, Schlunssen V, Isaksson M, Schmidt SAJ, Kolstad HA. Prevalence of skin sensitization and dermatitis among epoxy-exposed workers in the wind turbine industry. Br J Dermatol. 2022 Dec;187(6):988-996. doi: 10.1111/bjd.21830. Epub 2022 Sep 16. PMID 35972390
- [Background] Ponten A, Carstensen O, Rasmussen K, Gruvberger B, Isaksson M, Bruze M. Epoxy-based production of wind turbine rotor blades: occupational contact allergies. Dermatitis. 2004 Mar;15(1):33-40. doi: 10.2310/6620.2004.20433. PMID 15573646